CLINICAL TRIAL: NCT06367660
Title: Comparison Between Hyperbaric Bupivacaine With Fentanyl vs. Hyperbaric Bupivacaine With Dexmedetomidine in Reducing Visceral Pain During Cesarean Delivery Under Spinal Anaesthesia: A Prospective Randomised Double-Blind Study
Brief Title: Comparison Between Hyperbaric Bupivacaine With Fentanyl vs. Hyperbaric Bupivacaine With Dexmedetomidine in Reducing Visceral Pain During Cesarean Delivery Under Spinal Anaesthesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Sujan Dhakal, MD, Consultant Anaesthesiologist, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 98-2024
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Visceral Pain
MeSH Terms: conditions — Visceral Pain

STUDY DESIGN:
Intervention Model Description: Research method: Quantitative Type of study: Randomized, interventional, comparative study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine with Fentanyl (BF) (Active Comparator): In patients undergoing elective LSCS under subarachnoid block, group BF will receive 0.5% hyperbaric bupivacaine 10mg (2ml) with fentanyl 10 mcg (0.2ml) with total of 2.2 ml . Assessment of intraoperative visceral pain will be done by self-reporting of patients, who are previously educated, as poorly localized discomfort or dragging, pulling heaviness or unpleasant feeling or pain with or without nausea and will be categorized according to preformed scale.
  Interventions: Drug: Intrathecal Bupivacaine-Fentanyl and Bupivacaine-Dexmedetomidine
- Bupivacaine with Dexmedetomidine (BD) (Active Comparator): In patients undergoing elective LSCS under subarachnoid block, group BD will receive 0.5% hyperbaric bupivacaine 10 mg with Dexmedetomidine 5mcg (0.2ml) total volume 2.2ml. Assessment of intraoperative visceral pain will be done by self-reporting of patients, who are previously educated, as poorly localized discomfort or dragging, pulling heaviness or unpleasant feeling or pain with or without nausea and will be categorized according to preformed scale.
  Interventions: Drug: Intrathecal Bupivacaine-Fentanyl and Bupivacaine-Dexmedetomidine

INTERVENTIONS:
Drug: Intrathecal Bupivacaine-Fentanyl and Bupivacaine-Dexmedetomidine — In patients undergoing elective LSCS under subarachnoid block, group BF will receive 0.5% hyperbaric bupivacaine 10mg (2ml) with fentanyl 10 mcg (0.2ml) with total of 2.2 ml and group BD will receive 0.5% hyperbaric bupivacaine 10 mg with Dexmedetomidine 5mcg (0.2ml) total volume 2.2ml. Assessment of intraoperative visceral pain will be done by self-reporting of patients, who are previously educated, as poorly localized discomfort or dragging, pulling heaviness or unpleasant feeling or pain with or without nausea and will be categorized according to preformed scale.

SUMMARY:
In patients undergoing elective LSCS under subarachnoid block, group BF will receive 0.5% hyperbaric bupivacaine 10mg (2ml) with fentanyl 10 mcg (0.2ml) with total of 2.2 ml and group BD will receive 0.5% hyperbaric bupivacaine 10 mg with Dexmedetomidine 5mcg (0.2ml) total volume 2.2ml. Assessment of intraoperative visceral pain will be done by self-reporting of patients, who are previously educated, as poorly localized discomfort or dragging, pulling heaviness or unpleasant feeling or pain with or without nausea and will be categorized according to preformed scale

DETAILED DESCRIPTION:
Hours prior to surgery

* All the patients included in the study will be explained in detail about the purpose of the study, need, benefits and risks of procedure.
* They will be instructed on the method used for sensory and motor assessments.
* In addition, they will be explained about numerical rating scale of pain, how to use it and rate it and about symptoms of the visceral pain (if any) during SAB in intraoperative period.
* Written informed consent will be obtained during pre-anaesthetic check-up.
* Fasting period will be ensured before taking to pre-operative room.
* Premedication will be done with Tab. Pantoprazole 40 mg and Tab. Metoclopramide 10 mg at 10 pm the day before surgery and 6 am in morning of surgery will be ensured.

Before surgery

* In pre-operative room, a peripheral intravenous (IV) line will be established with 18-G IV cannula.
* Preloading will be done with 10 ml/kg of Lactated Ringer's solution.
* Baseline blood pressure, mean arterial pressure, heart rate, respiratory rate, SpO2, fetal heart rate will be recorded in pre-delivery room.

In the operation theater:

* Standard monitor including electrocardiography, non-invasive blood pressure monitoring and pulse oximetry will be attached.
* Patient will be positioned in sitting position.
* Painting of the patient's back with 10% Povidine Iodine and draping with sterile drapes will be done.
* Identification of intervertebral space will be done by noting the location of the L4 spinous process on Tuffier's line (line connecting the highest point of the iliac crests).
* Under all aseptic precautions, the skin will be infiltrated with lidocaine 2%, then a 25-gauge Quincke's spinal needle (Spinocan, B Braun medical Industries, Malaysia) will be introduced at L3-L4 or L4-L5 intervertebral space using a midline approach in sitting position.
* After ensuring free flow of cerebrospinal fluid, study drug will be given over 12 - 15 sec.
* Study drugs would be prepared as follow In group BD, 0.5% hyperbaric bupivacaine (ANAWIN heavy, Neon Laborotaries, India) 10mg (2ml) with addition of 5 mcg (0.2ml) Dexmedetomidine (DEXTOMID, Neon Laborotaries, India) with total volume of 2.2 ml will be prepared.

In group BF, 0.5% hyperbaric bupivacaine (ANAWIN heavy, Neon Laborotaries, India) 10 mg (2ml) with addition of 10mcg (0.2ml) fentanyl (TROFENTYL, Troikaa pharmaceuticals, India) with total volume of 2.2 ml will be prepared.

* Immediately after administration of spinal anesthesia, patient will be positioned supine with wedge under right hip and the time will be recorded as "time-zero".
* Fetal heart rates will be noted for any bradycardia.
* Patients will receive oxygen 3L/min via nasal cannula if SpO2 decreases to <95 %
* NIBP and HR will be assessed every 3-minute following SAB for 15 minutes or until delivery of baby and thereafter every 5 minutes till the end of surgery.
* SpO2 and ECG were monitored continuously throughout the study period.
* Hypotension will be promptly treated with intravenous fluid bolus (200 ml) and Inj. Mephentermine 6mg IV boluses, which will be repeated if necessary.
* If bolus dose of Mephentermine exceeds 30mg then Inj. Phenylephrine 50 mcg IV will be given.
* Inj. Atropine 0.6mg will be given if bradycardia occurs.
* If respiratory depression occurs, it will be recorded and managed as:

RR ≤10 breaths /min physical stimulus will be given (tapping a patient's shoulder with calling her name) If RR is still not increased or RR less than or equal to 8 breaths /min Inj Naloxone 0.4 mg IV will be given and will be repeated after 2-3 min if necessary. Dose of Naloxone will not be exceeded 10mg/ day.

* Sensory level will be assessed bilaterally along the mid clavicular line using spirit-soaked cotton until block reached upto T6 dermatome and time will be noted.
* Motor block will be assessed based on Modified Bromage Scale and time will be noted.
* Surgery will be allowed as soon as upper sensory level reaches T6 and Bromage scale of M3.
* Thereafter, the level will be checked every 2 min until maximal sensory block level is confirmed.
* Intra operative pain will be assessed whenever the patient complains of pain or discomfort during surgery.
* If somatic pain occurs (at time of incision to skin or subcutaneous tissue), spinal anesthesia will be converted to general anesthesia and excluded from study.
* Whenever visceral pain occur, participants were encouraged to self-report such experience and were enquired every five minutes interval during surgery. For analysis, visceral pain outcome, was categorized as following:6

  1. Excellent, no complaints,
  2. Mild discomfort, requiring no analgesic,
  3. Intermediate discomfort accompanied by nausea requiring anti-emetic,
  4. Severe discomfort accompanied by pain requiring analgesic, and
  5. Failed SA, requiring GA.
* Assessment of visceral pain will be mainly done during; Delivery of baby with fundal pressure application: when pulling out the head of baby from uterus Exteriorization of uterus: temporary extraction of uterus outside the abdominal cavity to facilitate uterine incision repair Handling of other intraperitoneal organs like bowels, adenexa so as to clear off the secretions and blood Suturing of visceral peritoneum Placement of uterus back to abdominal cavity after repair
* The occurrence of nausea was correlated with the decrement of SBP and/or HR and addressed first.
* Nausea-vomiting occurring otherwise was treated with Ondansetron, Metoclopramide, and Dexamethasone as needed.
* Anxiety was addressed with Midazolam (maximum three mg).
* Each time NRS is 4 or more it will be considered as inadequate analgesia7, and inj. Fentanyl 25 mcg will be given IV bolus.
* We will wait for 3 min for its adequate effect.
* If still pain persists, then the dose of fentanyl will be increased to 1 mcg/kg.
* After 2 doses of fentanyl, if pain still persists then Inj. Ketamine 0.5mcg/kg IV will be given.
* If still pain is unbearable, general anesthesia will be administered.
* The need to convert to GA will be noted.
* Level of consciousness will be measured using sedation scale (POSS scale)8
* Incidence of shivering will be noted during intraoperative period, where temperature of OR will be kept between 18-21 degree Celsius.
* Occurrence of side effects such as nausea, vomiting, dizziness, pruritus, bradycardia, decrease in SPO2 and respiratory rate will be recorded and treated according to severity.
* Any patients who will have these sign and symptoms will be assessed every 15 min in OR and recovery room.
* Following delivery of the baby, Inj. oxytocin 3 IU will be administered bolus.
* Continuous infusion of oxytocin drip will be given as per need after communicating with obstetrician
* APGAR score of the neonate will be evaluated at 1 minute and 5 minutes.
* Weight of baby will be noted.
* Postoperatively, patients will be monitored hourly for hemodynamic changes and for any side effects of study drugs upto 6hrs.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean deliveries under SAB
* ASA PS II
* Age ≥18 years
* Term pregnancy ≥37 weeks of gestation
* Height ≥ 150

Exclusion Criteria:

* Patients with medical disorder in pregnancy (neurological, psychiatric, cardiopulmonary,
* hepatorenal diseases, coagulopathy)
* Patient refusal to participate
* Allergy or hypersensitivity to LA, fentanyl or dexmedetomidine
* Patients with communication problem
* Patient with bradycardia (HR- less than 60)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant female planned for elective C-section
Enrollment: 168 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | Intraoperative
  To compare the incidence of intraoperative visceral pain between participants of two groups.

SECONDARY OUTCOMES:
Secondary Outcome | Intraoperative
  To compare occurrence of intraoperative shivering between participants of two groups.
  To compare the intraoperative systolic blood pressure, diastolic blood pressure, mean arterial pressure and heart rate between two groups To compare the incidence of side effects like nausea, vomiting, respiratory depression, pruritus, between two groups To compare the neonatal APGAR score between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Sujan Dhakal, Principal Investigator — Ministry of health and population

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhakal S, Shrestha M, Gautam E, Suwal A, Dhakal S, Dhakal S. Comparison of hyperbaric bupivacaine with fentanyl vs. hyperbaric bupivacaine with dexmedetomidine in reducing visceral pain during cesarean delivery under spinal anesthesia: study protocol. Pain Manag. 2025 Oct;15(10):651-658. doi: 10.1080/17581869.2025.2543232. Epub 2025 Aug 6. PMID 40765391